CLINICAL TRIAL: NCT02544815
Title: Assessment of the Efficacy and Safety of a Short Term Treatment With Digoxin on Patients With Acute Heart Failure Syndromes. A Randomized Controlled Trial.
Brief Title: Digoxin Short Term Treatment Assessment Randomized Trial in AHF
Acronym: DIG-STA-AHF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Digoxin - START - AHF
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Acute Heart Failure
Keywords: digoxin, eficacy, safety
MeSH Terms: interventions — Digoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digoxin (Active Comparator): Oral digoxin 0.25 mg: one pill per day for 30 consecutive days.
  Interventions: Drug: Digoxin
- Placebo (Placebo Comparator): Oral placebo for 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Digoxin — Digoxin 0.25 mg pills
  Arms: Digoxin
Drug: Placebo — Placebo pills
  Arms: Placebo

SUMMARY:
AHFS management is challenging and most of the used drugs has failed to decrease post-discharge mortality and readmission rates which represent the most important goal in AHFS.

Digoxin processes many characteristics of a beneficial drug for heart failure, however recent publications has rose concerns about its safety profile and therefore decreasing its use.

Whether digoxin is efficient and safe in short term treatment of acute heart failure is a question that should be studied.

DETAILED DESCRIPTION:
AHFS management is challenging given the heterogeniety of the patient population, absence of a universally accepted definition, incomplete understanding of its pathophysiology, and lack of evidence based guidelines.

The majority of patients appear to respond well to initial therapies consisting of loop diuretics and vasoactive agents. however, this treatments failed to decrease post-discharge mortality and readmission rates which represent the most important goal in AHFS.

In the last few years, many drugs has been tested in AHFS setting trying to adress this issue, however results has been disappointing in term of efficacy and / or safety.

Although evidence supports the beneficial effects of digoxin on hemodynamic, neurohormonal, and electrophysiological parameters in patients with CHF, recent publications has rose concerns about its safety profile and therefore decreasing its use.

The effects of digoxin alone or in combination with other vasodilators are seen within few hours of its administration and result in increased cardiac output, decreased pulmonary wedge pressure, increased ejection fraction, and improved neurohormonal profile without changes in blood pressure.

All this findings made us rose the question of whether digoxin is effective or not in short term treatment of acute heart failure ? Additionnel treatments for AHF were given according left to ACCF/AHA for the managementof heart failure .

Blood testing for scanner digoxin magerments will be confirmed at H8, h24 and H72 after the post protocol treatment admession treatment administration.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed written consent.
* Male or female aged ≥18 years old.
* Admitted for acute heart failure defined by the presence of dypnea at rest or with minimal exertion , pulmonary congestion on chest radiograph ; and increased natriutic peptide concentrations ( BNP >=350 pg/ml) or NTproBNP >=1400 pg/ml ) .
* Able to be randomized within 12 hours from presentation to the hospital.

Exclusion Criteria:

* Pregnant or breast feeding women.
* Known severe or terminal renal failure.
* Previous hepatic impairment.
* Major surgery within 30 days.
* Hematocrit < 25%.
* Alteration of consciousness GCS < 15
* Critically ill patients needing immediate mechanical hemodynamic of ventilatory support.
* Confirmed or suspected diagnosis of ACS within 45 days before inclusion.
* Severe arrhythmias including significant sinoatrial or atrioventricular blocks or WPW syndrome.
* Implantable cardiac devices including pacemakers and defibrillators.
* Hypertrophic obstructive, restrictive, or constrictive cardiomyopathy.
* Noncardiac pulmonary edema, including suspected sepsis.
* Severe pulmonary disease
* Significant stenotic valvular disease .
* Hyperkalemia > 5.5 mmol /L .
* Administration of an investigational drug or implantation of an investigational device or participation in another trial within 30 days before screening.
* Previous treatment with digoxin within 15 days before inclusion or contra-indications to digoxin.
* Inability to follow instructions or comply with follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
30 days mortality and rehospitalization rate | 30 days

SECONDARY OUTCOMES:
Hemodynamic improvement | 3 days
  Change in hemodynamic parameters as quantified by the area under the curve of bio-impedance thoracic fluid contenant (TFC), lung ultrasound (LUS) congestion score and BNP serum levels, from baseline to day 3.
Need for hospitalization | 3 days
Length of stay in hospital | from baseline to hospital discharge
AUC of dyspnea VAS scores | 3 days
  Change in patient-reported dyspnea as quantified by the area under the curve (AUC) of visual analogue scale (VAS) scores (0-100 mm scale) : a dyspnea VAS score of 0 corresponds to the patient's subjective feeling of "I Can Breathe Normally" and a dyspnea VAS score of 100 corresponds to "I Can't Breathe At All.
Improvement of patient-reported dyspnea | [Time Frame: 6, 12, and 24 hours from start of the study medication]
  Improvement of patient-reported dyspnea relative to the start of study drug using a 5 point likert scale at 6, 12, and 24 hours, where a responder was a patient with better or markedly betted dyspnea at all three of those time points.
Dyspnea resolution time | 3 days
  defined as the time between the start of study drug and the reduction of at least 50% of the dyspnea VAS score from baseline.
Digoxin related adverse events | 30 days
  Occurrence of major adverse events related to digoxin and implicating its discontinuation.
  Admitted major side effects of digoxin are: Severe ventricular arrhythmias including ventricular tachycardia or fibrillation, Severe bradycardia, Second- or third-degree heart block not responsive to atropine, Serum potassium levels exceeding 5.5 mEq/L with rapidly progressive signs and symptoms of digoxin toxicity, Neurologic symptoms (eg, visual disturbances, disorientation, and confusion).
Worsening renal function | 30 days
  worsening renal function under treatment is defined as a relative increase in serum creatinine of at least 25% from baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University Hospital of Monastir
Locations (2):
- Tunisia (2):
  - Sahloul University Hospital, Hammam Sousse, Sousse Governorate
  - Fattouma Bourguiba University Hospital, Monastir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gheorghiade M, Zannad F, Sopko G, Klein L, Pina IL, Konstam MA, Massie BM, Roland E, Targum S, Collins SP, Filippatos G, Tavazzi L; International Working Group on Acute Heart Failure Syndromes. Acute heart failure syndromes: current state and framework for future research. Circulation. 2005 Dec 20;112(25):3958-68. doi: 10.1161/CIRCULATIONAHA.105.590091. No abstract available. PMID 16365214
- [Background] Digitalis Investigation Group. The effect of digoxin on mortality and morbidity in patients with heart failure. N Engl J Med. 1997 Feb 20;336(8):525-33. doi: 10.1056/NEJM199702203360801. PMID 9036306
- [Background] Hashim T, Elbaz S, Patel K, Morgan CJ, Fonarow GC, Fleg JL, McGwin G, Cutter GR, Allman RM, Prabhu SD, Zile MR, Bourge RC, Ahmed A. Digoxin and 30-day all-cause hospital admission in older patients with chronic diastolic heart failure. Am J Med. 2014 Feb;127(2):132-9. doi: 10.1016/j.amjmed.2013.08.006. Epub 2013 Sep 23. PMID 24067296